CLINICAL TRIAL: NCT00718029
Title: MK: Raltegravir Concentrations in Cerebrospinal Fluid
Brief Title: Cerebrospinal Fluid (CSF) Raltegravir Substudy
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MK: 33132
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus; Cerebrospinal Fluid; Raltegravir; Drug Concentrations
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CSF, PBMC, plasma

SUMMARY:
The purpose of this study is to measure concentrations of Raltegravir in cerebrospinal fluid.

The hypotheses are:

* Raltegravir concentrations in CSF will be measurable
* Raltegravir concentrations in CSF will remain constant, while plasma concentrations vary widely leading to highly variable CSF-to-plasma ratios.
* Following at least 4 weeks of Raltegravir-containing combination therapy, HIV RNA levels in CSF will be below 50 copies/mL in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in a raltegravir parent protocol at UCSD.
* Willing to undergo lumbar puncture.
* Able to give informed consent. If cognitively impaired, a test will be administered to ensure adequate comprehension of the consent document and procedure.

Exclusion Criteria:

* Relative or absolute contraindication to lumbar puncture, such as current coagulopathy, thrombocytopenia (platelets<50,000/µL), hemophilia, or use of anticoagulant medication.
* Psychiatric disease that would interfere with study participation, in the opinion of the investigator.
* No major opportunistic infections within 30 days.
* Moderate or severe cognitive impairment. The proposed study does not have a neuropsychological objective.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected from participants already enrolled in Merck-sponsored Raltegravir Clinical Trials.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Letendre, MD, Principal Investigator — University of California, San Diego AntiViral Research Center